CLINICAL TRIAL: NCT01564368
Title: Diffusion Weighted MR Imaging Biomarkers for Assessment of Breast Cancer Response to Neoadjuvant Treatment: A Sub-study of the I-SPY 2 TRIAL (Investigation of Serial Studies to Predict Your Therapeutic Response With Imaging And MoLecular Analysis)
Brief Title: DWI in Assessing Treatment Response in Patients With Breast Cancer Receiving Neoadjuvant Chemotherapy
Acronym: ACRIN6698
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000729174; ACRIN-6698 (Other: NCI CIP); U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2012-03-24; First posted 2012-03-27 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; HER2-negative breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diffusion Weighted-MRI (Experimental): Participants on all arms of the I-SPY II trial will undergo diffusion-weighted magnetic resonance imaging as described in the ACRIN 6698 protocol. The experimental component/intervention is whether DW-MRI can predict therapeutic response in neoadjuvant treatment for breast cancer.
  Interventions: Procedure: diffusion-weighted magnetic resonance imaging

INTERVENTIONS:
Procedure: diffusion-weighted magnetic resonance imaging — diffusion-weighted magnetic resonance imaging examination and subsequent radiologist interpretation
  Other Names: functional MRI; DWI; diffusion-weighted MRI; DW-MRI

SUMMARY:
RATIONALE: Imaging procedures, such as diffusion-weighted magnetic resonance imaging (DWI) and dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI), may help in evaluating how well patients with breast cancer respond to treatment.

PURPOSE: This research trial studies DWI and DCE-MRI in assessing treatment response in patients with breast cancer undergoing neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if the change in tumor apparent diffusion coefficient (ADC) value measured from each treatment timepoint to baseline is predictive of pathologic complete response (pCR).

Secondary

* To determine if the combined measurement of change in tumor ADC value, change in tumor volume, and change in peak signal-enhancement ratio (SER) is predictive of pCR.
* To investigate the relative effectiveness of the individual measurements, change in tumor ADC value, change in tumor volume, and change in peak SER for predicting pCR in experimental treatment arms.
* To assess the test-retest reproducibility of ADC metrics applied to breast tumors.

OUTLINE: This is a multicenter study.

Patients undergo diffusion-weighted magnetic resonance imaging (DWI) at baseline, after week 3 of neoadjuvant paclitaxel regimen, and prior to and after completion of 4 courses of neoadjuvant chemotherapy. Patients then undergo surgery. Patients undergo DWI prior to contrast administration for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI).

After completion of treatment procedure, patients are followed up for 5 years on the I-SPY 2 TRIAL.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets I-SPY 2 TRIAL inclusion criteria

  * High-risk for recurrent disease

PATIENT CHARACTERISTICS:

* Able to tolerate imaging required by protocol

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2012-08-27 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nola M. Hylton, PhD, Principal Investigator — University of California, San Francisco
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - University of Washington/SCCA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
See ACRIN data sharing Policy https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx
Supporting Information: Study Protocol, SAP
Time Frame: 6mo post publication
Access Criteria: upon request
URL: https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx

REFERENCES:
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132
- [Result] Li W, Partridge SC, Newitt DC, Steingrimsson J, Marques HS, Bolan PJ, Hirano M, Bearce BA, Kalpathy-Cramer J, Boss MA, Teng X, Zhang J, Cai J, Kontos D, Cohen EA, Mankowski WC, Liu M, Ha R, Pellicer-Valero OJ, Maier-Hein K, Rabinovici-Cohen S, Tlusty T, Ozery-Flato M, Parekh VS, Jacobs MA, Yan R, Sung K, Kazerouni AS, DiCarlo JC, Yankeelov TE, Chenevert TL, Hylton NM. Breast Multiparametric MRI for Prediction of Neoadjuvant Chemotherapy Response in Breast Cancer: The BMMR2 Challenge. Radiol Imaging Cancer. 2024 Jan;6(1):e230033. doi: 10.1148/rycan.230033. PMID 38180338
- [Result] Partridge SC, Zhang Z, Newitt DC, Gibbs JE, Chenevert TL, Rosen MA, Bolan PJ, Marques HS, Romanoff J, Cimino L, Joe BN, Umphrey HR, Ojeda-Fournier H, Dogan B, Oh K, Abe H, Drukteinis JS, Esserman LJ, Hylton NM; ACRIN 6698 Trial Team and I-SPY 2 Trial Investigators. Diffusion-weighted MRI Findings Predict Pathologic Response in Neoadjuvant Treatment of Breast Cancer: The ACRIN 6698 Multicenter Trial. Radiology. 2018 Dec;289(3):618-627. doi: 10.1148/radiol.2018180273. Epub 2018 Sep 4. PMID 30179110
- [Result] Newitt DC, Amouzandeh G, Partridge SC, Marques HS, Herman BA, Ross BD, Hylton NM, Chenevert TL, Malyarenko DI. Repeatability and Reproducibility of ADC Histogram Metrics from the ACRIN 6698 Breast Cancer Therapy Response Trial. Tomography. 2020 Jun;6(2):177-185. doi: 10.18383/j.tom.2020.00008. PMID 32548294
- [Result] Newitt DC, Zhang Z, Gibbs JE, Partridge SC, Chenevert TL, Rosen MA, Bolan PJ, Marques HS, Aliu S, Li W, Cimino L, Joe BN, Umphrey H, Ojeda-Fournier H, Dogan B, Oh K, Abe H, Drukteinis J, Esserman LJ, Hylton NM; ACRIN Trial Team and I-SPY 2 TRIAL Investigators. Test-retest repeatability and reproducibility of ADC measures by breast DWI: Results from the ACRIN 6698 trial. J Magn Reson Imaging. 2019 Jun;49(6):1617-1628. doi: 10.1002/jmri.26539. Epub 2018 Oct 22. PMID 30350329
- [Result] Partridge SC, Steingrimsson J, Newitt DC, Gibbs JE, Marques HS, Bolan PJ, Boss MA, Chenevert TL, Rosen MA, Hylton NM. Impact of Alternate b-Value Combinations and Metrics on the Predictive Performance and Repeatability of Diffusion-Weighted MRI in Breast Cancer Treatment: Results from the ECOG-ACRIN A6698 Trial. Tomography. 2022 Mar 4;8(2):701-717. doi: 10.3390/tomography8020058. PMID 35314635
- [Result] Newitt DC, Tan ET, Wilmes LJ, Chenevert TL, Kornak J, Marinelli L, Hylton N. Gradient nonlinearity correction to improve apparent diffusion coefficient accuracy and standardization in the american college of radiology imaging network 6698 breast cancer trial. J Magn Reson Imaging. 2015 Oct;42(4):908-19. doi: 10.1002/jmri.24883. Epub 2015 Mar 11. PMID 25758543
- See also: National Cancer Institute's Clinical trial database — https://clinicaltrials.gov/ct2/show/NCT01564368

RESULTS

PARTICIPANT FLOW:
Groups:
- Diffusion Weighted-MRI: Participants on all arms of the I-SPY II trial will undergo diffusion-weighted magnetic resonance imaging as described in the ACRIN 6698 protocol. The experimental component/intervention is whether DW-MRI can predict therapeutic response (pathological Complete Response: pCR) in neoadjuvant treatment for breast cancer.
Period: Overall Study
Arm/Group | Diffusion Weighted-MRI
Started | 406
Randomized in Parent Study | 272
Acceptable Baseline Imaging | 263
Acceptable Post Baseline Image | 242
Baseline and Early Treatment Usable | 227
Baseline and Mid-treatment Usable | 210
Baseline and Post-Treatment Usable | 186
Usable Re-test Scan | 71
Completed | 242
Not Completed | 164
Not completed — Ineligible | 18
Not completed — Not Randomized in Parent study | 116
Not completed — Baseline Imaging failed QC requirements | 9
Not completed — No Acceptable post-baseline imaging | 21

BASELINE CHARACTERISTICS:
Population: Eligible randomized participants with a usable Baseline DWI-MRI and at least 1 other usable DWI scan at early-treatment, late-treatment, or pre-surgery
Groups:
- Diffusion Weighted-MRI: Participants on all arms of the I-SPY II trial with both a diffusion-weighted magnetic resonance imaging (DWI-MRI) scan at baseline and 1 post-baseline timepoint (early-treatment, mid-treatment, or post-treatment). The experimental component/intervention is whether DW-MRI can predict therapeutic response in women receiving neoadjuvant treatment for breast cancer.
Arm/Group | Diffusion Weighted-MRI
Number analyzed (Participants) | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (10.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 154
  Unknown or Not Reported | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 26
  White | 173
  More than one race | 0
  Unknown or Not Reported | 26

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR)
Description: Pathologic complete response (pCR) is defined as the lack of all signs of cancer in tissue samples removed during surgery after Neoadjuvant treatment for Breast cancer.
  ie., no residual invasive disease in either breast or axillary lymph nodes after neoadjuvant therapy (ypT0/is, ypN0) Histopathologic analysis was performed using the Residual Cancer Burden system
Time Frame: Surgery
Measure: Count of Participants; unit: Participants
Groups:
- Early Treatment Change: Participants who had both the pre-treatment (baseline) and the early-treatment (after 3 weekly doses of paclitaxel/taxane-based therapy) scans
- Mid-Treatment Change: Participants who had both the pre-treatment (baseline) and the mid-treatment (after 12 weeks, between taxane and anthracycline regimens) scans
- Post-Treatment Change: Participants who had both the pre-treatment (baseline) and the post-treatment (post-treatment after all chemotherapy, prior to surgery) scans
Arm/Group | Early Treatment Change | Mid-Treatment Change | Post-Treatment Change
Number analyzed (Participants) | 227 | 210 | 186
Participants
  Pathological Complete Responders (pCR) | 71 | 70 | 63
  Non-Responders(pCR-) | 156 | 140 | 123
Statistical Analysis 1: Comparison: Early Treatment Change; Receiver Operating Characteristic curves and the corresponding Area Under the Curve (AUC), were estimated for the change in Apparent Diffusion Coefficients (ADC1 - ADC0)/ADC0 (Test: %change in ADC; Reference: pCR) detect a difference of 0.15 between the AUC under H0: AUC=0.5 and an AUC under the alternative hypothesis of 0.65. It was assumed that the number of pCR non-responders would be approximately 2.7 times greater than the number of complete responders; Test type: Superiority; p = 0.484, Z-test — Bonferroni's correction was used for multiple comparisons adjustment, where p<0.003 (0.05/15) was considered statistically significant; The empirical AUC was tested by using variance derived from the method of DeLong; area under the curve (AUC) = 0.53, 95% CI 1-sided [upper limit 0.61] — Receiver operating characteristic curve and AUC were estimated empirically, and its 95% CI was constructed using variance derived from DeLong's method
Statistical Analysis 2: Comparison: Mid-Treatment Change; Receiver Operating Characteristic curves and the corresponding Area Under the Curve (AUC), were estimated for the change in Apparent Diffusion Coefficients (ADC2 - ADC0)/ADC0 (Test: %change in ADC; Reference: pCR) detect a difference of 0.15 between the AUC under H0: AUC=0.5 and an AUC under the alternative hypothesis of 0.65. It was assumed that the number of pCR non-responders would be approximately 2.7 times greater than the number of complete responders; Test type: Superiority; p = 0.017, Z-test — [p-value comment as in outcome 1, analysis 1]; The empirical AUC was tested by using variance derived from the method of DeLong; area under the curve = 0.60, 95% CI 1-sided [upper limit 0.68] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Post-Treatment Change; Receiver Operating Characteristic curves and the corresponding Area Under the Curve (AUC), were estimated for the change in Apparent Diffusion Coefficients (ADC3 - ADC0)/ADC0 (Test: %change in ADC; Reference: pCR) detect a difference of 0.15 between the AUC under H0: AUC=0.5 and an AUC under the alternative hypothesis of 0.65. It was assumed that the number of pCR non-responders would be approximately 2.7 times greater than the number of complete responders; Test type: Superiority; p = 0.013, Z-test — Bonferroni's correction was used for multiple comparisons adjustment, where p<0.003 (0.05/15) is considered statistically significant; The empirical AUC was tested by using variance derived from the method of DeLong; area under the curve = 0.61, 95% CI 1-sided [upper limit 0.69] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Functional Tumor Volume (FTV) as a Predictor of Pathologic Complete Response (pCR)
Description: Pathologic complete response (pCR) is defined as the lack of all signs of cancer in tissue samples removed during surgery after Neoadjuvant treatment for Breast cancer.
  ie., no residual invasive disease in either breast or axillary lymph nodes after neoadjuvant therapy (ypT0/is, ypN0) Histopathologic analysis was performed using the Residual Cancer Burden system Functional tumor volume (FTV) (units cm3) was computed by summing all tumor voxels meeting specific enhancement criteria, with customized thresholds for each site to account for variability in MR imaging systems
Time Frame: Surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment Change | Mid-Treatment Change | Post-Treatment Change
Number analyzed (Participants) | 227 | 210 | 186
Participants
  Pathological Complete Responders (pCR) | 71 | 70 | 63
  Non-Responders(pCR-) | 156 | 140 | 123
Statistical Analysis 1: Comparison: Early Treatment Change; Receiver Operating Characteristic curves and the corresponding Area Under the Curve (AUC), were estimated for the change in functional tumor volumes (FTV1 - FTV0)/FTV0 (Test: %change in FTV; Reference: pCR) detect a difference of 0.15 between the AUC under H0: AUC=0.5 and an AUC under the alternative hypothesis of 0.65. It was assumed that the number of pCR non-responders would be approximately 2.7 times greater than the number of complete responders; Test type: Superiority; p < 0.001, Z-test — [p-value comment as in outcome 1, analysis 1]; The empirical AUC was tested by using variance derived from the method of DeLong; area under the curve = 0.68, 95% CI 1-sided [upper limit 0.75] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mid-Treatment Change; Receiver Operating Characteristic curves and the corresponding Area Under the Curve (AUC), were estimated for the change in functional tumor volumes (FTV2 - FTV0)/FTV0 (Test: %change in FTV; Reference: pCR) detect a difference of 0.15 between the AUC under H0: AUC=0.5 and an AUC under the alternative hypothesis of 0.65. It was assumed that the number of pCR non-responders would be approximately 2.7 times greater than the number of complete responders; Test type: Superiority; p < 0.001, Z-test — [p-value comment as in outcome 1, analysis 1]; The empirical AUC was tested by using variance derived from the method of DeLong; area under the curve = 0.63, 95% CI 1-sided [upper limit 0.71] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Post-Treatment Change; Receiver Operating Characteristic curves and the corresponding Area Under the Curve (AUC), were estimated for the change in functional tumor volumes (FTV3 - FTV0)/FTV0 (Test: %change in FTV; Reference: pCR) detect a difference of 0.15 between the AUC under H0: AUC=0.5 and an AUC under the alternative hypothesis of 0.65. It was assumed that the number of pCR non-responders would be approximately 2.7 times greater than the number of complete responders; Test type: Superiority; p < 0.001, Z-test — [p-value comment as in outcome 1, analysis 1]; The empirical AUC was tested by using variance derived from the method of DeLong; area under the curve = 0.68, 95% CI 1-sided [upper limit 0.75] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Determine the Accuracy of Predictive Models Including Covariates for Combined Measurement of Change in Tumor ADC Value, Change in Tumor Volume, and Other Variables
Description: Accuracy will be measured as the Area under the Receiver Operating Characteristic Curve (AUC) Predictive logistic regression modeling was performed in 207 patients with complete mid-treatment ΔADC and ΔFTV data.
  To build prediction models with ADC and other variables, a data-splitting approach was used where a randomly selected 60% of participants (124 patients), stratified according to pCR status and tumor subtype, were selected as the training data set and the rest (86 patients) as the test set. Logistic regression with backward variable selection was used to construct the prediction models, which were then applied to the remaining 40% of the data to obtain predictive scores for each participant.
Time Frame: baseline and mid-treatment
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Full Combined Model: The data were split into a 60% training set (124 patients, randomly selected and stratified according to tumor subtype) and a 40% validation set (86 patients). Characteristics of the 86-patient test set were representative of the full analysis set, A predictive model, combining ΔADC, ΔFTV, and cancer subtype, was used to predict performance
- Optimized Model: Backward selection was used to optimize the full model, and ΔFTV was eliminated, and the final prediction model retained ΔADC and tumor subtype as predictors.
- ΔADC Alone: Tumor ADC change (the percentage change from the pretreatment to mid-treatment (ΔADC)) as the sole predictor of pCR
Arm/Group | Full Combined Model | Optimized Model | ΔADC Alone
Number analyzed (Participants) | 86 | 86 | 86
probability | 0.71 [0.59 to 0.84] | 0.72 [0.61 to 0.83] | 0.57 [0.44 to 0.70]
Statistical Analysis 1: Comparison: Optimized Model vs ΔADC Alone; AUC (optimized) = AUC (ΔADC); Test type: Equivalence — no equivalence margin was used; p = 0.032, z-test

4. Secondary Outcome: Repeatability Coefficient (RC)Test-retest Metric for Reproducibility of ADC as Applied to Breast Tumors
Description: within-subject standard deviation (wSD) Repeatability coefficient (RC): [RC = 2.77*wSD] (units: 10E-3 mm/sec^2)
  Smaller values of RC, bounded [0, ...), represent agreement
Time Frame: baseline (pre-treatment) or after 3 weeks of taxane-based treatment (early-treatment)
Measure: Number (95% Confidence Interval); unit: 10E-3 mm/sec^2
Groups:
- Test-Retest Subjects: Test and retest DWI measurements for a given patient were performed on the same day in a single imaging session. The patient was positioned normally (prone) and scanned with initial localization, T2W, and DWI acquisitions (2017 QIBA Profile). A single test/retest study was conducted for each consented subjects at either T0 or T1, with T0 specified as the preferred timepoint.
Arm/Group | Test-Retest Subjects
Number analyzed (Participants) | 71
10E-3 mm/sec^2 | 0.16 [0.13 to 0.19]

5. Secondary Outcome: Within-subject Coefficient of Variation (wCV) Test-retest Metric for Reproducibility of ADC as Applied to Breast Tumors
Description: within-subject standard deviation (wSD) Within-subject coefficient of variation (wCV): [wCV = 100%*wSD/mean]
  Smaller values of wCV bounded for [0,...) represent better agreement
Time Frame: baseline (pre-treatment) or after 3 weeks of taxane-based treatment (early-treatment)
Measure: Number (95% Confidence Interval); unit: coefficient of variation
Arm/Group | Test-Retest Subjects
Number analyzed (Participants) | 71
coefficient of variation | 4.8 [4.0 to 5.7]

6. Secondary Outcome: ICC Test-retest Metric for Reproducibility of ADC as Applied to Breast Tumors
Description: Test and retest DWI measurements for a given patient were performed on the same day in a single imaging session.
  Intraclass correlation coefficient (ICC) is derived from the analysis of variance (ANOVA) model estimates (Barnhart,Haber, Lin 2007),
  Larger values of ICC (bounded [-1,1]) represent agreement
Time Frame: baseline (pre-treatment) or after 3 weeks of taxane-based treatment (early-treatment)
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Test-Retest Subjects
Number analyzed (Participants) | 71
correlation coefficient | 0.97 [0.95 to 0.98]

7. Secondary Outcome: Agreement Index (AI) Test-retest Metric for Reproducibility of ADC as Applied to Breast Tumors
Description: Test and retest DWI measurements for a given patient were performed on the same day in a single imaging session.
  Agreement index (AI): (Zhang, Wang, Duan - 2014) is based on the data's overall ranking. AI confidence intervals were obtained via bootstrap method Larger values AI (bounded [0.5,1]) represent agreement
Time Frame: baseline (pre-treatment) or after 3 weeks of taxane-based treatment (early-treatment)
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Test-Retest Subjects
Number analyzed (Participants) | 71
probability | 0.83 [0.76 to 0.87]

ADVERSE EVENTS:
Time Frame: From registration to surgery or off study, for events occurring within 30 days of each DW-MRI exam
Arm/Group | Diffusion Weighted-MRI
All-Cause Mortality (participants affected / at risk) | 0/406
Serious Adverse Events (participants affected / at risk) | 0/406
Other Adverse Events (participants affected / at risk) | 0/406

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT01564368/Prot_SAP_000.pdf